CLINICAL TRIAL: NCT02660541
Title: A Pilot Study to Compare Efficacy of Allevyn® Silver Dressing and Betafoam® in Patients With Wound of Acute Burn Injury
Brief Title: Burn Wound Management of Betafoam® and Allevyn® Ag
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTF15-KR-401
Record Dates: First submitted 2016-01-13; First posted 2016-01-21 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Acute Burn
Keywords: Dressing for burn wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Betafoam (Active Comparator): Brand name: Betafoam® This is a medicated device (dressing) consisting of 3% povidone iodine.
  Interventions: Device: Betafoam
- Allevyn Silver dressing (Active Comparator): Brand name: Allevyn® Silver
  Interventions: Device: Allevyn Silver Dressing

INTERVENTIONS:
Device: Betafoam — Comparison between 2 medical devices
  Arms: Betafoam
Device: Allevyn Silver Dressing — Comparison between 2 medical devices
  Arms: Allevyn Silver dressing

SUMMARY:
This is a randomized, controlled, multi-centre, open-label study.

A total of 40 patients will be enrolled in this study. Patients will be randomly assigned to Betafoam® or Allevyn® Silver dressing for burn wounds after acute burn injury.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 19 years
2. Subjects of second-degree burn who have acute partial thickness burn (superficial to deep partial thickness) via investigator's visible assessment
3. Burn total body surface area of <15% range based on Lund and Browder chart presenting at the emergency room within the first 3~5 days post-injury will be considered for inclusion in this study.

   (If more than one burn wound is present that meets the inclusion criteria, the largest one among wounds that size are between 10x10 ㎝ and 20x20㎝ will be preferred to select as the Target wound.)
4. Subjects who voluntarily sign the informed consent form

Exclusion Criteria:

1. Pregnant & lactating females
2. Known allergy to the dressing product including PVP-I
3. Known hyperthyroidism or other acute thyroid diseases
4. Subject with clinical infection who should be administered antibiotics continuously after enrolment
5. Subject has any condition(s) that seriously compromises the patient's ability to complete this study.
6. Subject has participated in interventional study utilizing an investigational drug within the previous 30 days
7. Subject has one or more medical condition(s), diabetes, including renal, hepatic, hematologic, neurologic, or immune disease that presumably to hinder the wound healing processes by the physician's judgement.
8. Subjects who are immune suppressed states, under chemo- or radiotherapy.
9. The surgeon decides that surgery is necessary or requiring skin grafting.
10. Burn injury sites at the ends of extremities and genitalia
11. Burn injury caused of electronic burn
12. Subjects who have inhaled damage, severe head injury or fracture on burn wound
13. Scintillation scan for the diagnosis of thyroid takes at intervals of 1 to 2 weeks when using this dressing
14. Vulnerable subjects.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Comparison between Betafoam® and Allevyn® Silver dressing, measured by days needed for complete re-epithelialization in burn wounds | 28 days

SECONDARY OUTCOMES:
Safety assessed by documentation of adverse events, clinical laboratory results and vital signs | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Dohern Kim, Dr., Principal Investigator — Hangang Sacred Heart Hospital
Locations (1):
- Hallym University Hangang Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided